CLINICAL TRIAL: NCT03084367
Title: DEFINE PCI: Physiologic Assessment of Coronary Stenosis Following PCI
Brief Title: Physiologic Assessment of Coronary Stenosis Following PCI
Acronym: DEFINE PCI
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Collaborators: Duke Clinical Research Institute (Other); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 160101
Record Dates: First submitted 2017-03-13; First posted 2017-03-20 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Angina, Unstable; Angina, Stable
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Angina, Unstable; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iFR post angiographically successful PCI
  Interventions: Diagnostic Test: iFR pullback

INTERVENTIONS:
Diagnostic Test: iFR pullback — iFR pullback assessment post angiographically successful PCI

SUMMARY:
This is a pilot study designed to assess the relationship between iFR (instantaneous wave-free ratio) pullback and the distribution of coronary atheroma/stenoses as assessed by Quantitative Coronary Angiography (QCA) post angiographically successful PCI (Percutaneous Coronary Intervention).

DETAILED DESCRIPTION:
DEFINE-PCI is a multi-center, prospective, non-significant risk study in up to 25 centers in USA and internationally. Consented subjects with CAD (Coronary Artery Disease) who undergo physiologic lesion assessment with iFR<0.90 in at least 1 coronary artery are eligible for participation. After successful PCI to all culprit lesions based on angiographic assessment of the treating physician, a blinded post-PCI iFR and iFR pullback will be performed. The proportion of patients with impaired post-PCI iFR will be assessed, and the number of patients in whom ischemia could theoretically be normalized with further PCI determined. Additionally, the association between the post-PCI iFR results and cardiovascular events and clinical symptoms will be assessed. Follow-up will be at 1, 6 and 12 months, including administration of quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be > 18 years old
2. Subjects presenting with stable angina, silent ischemia or non-ST-elevation ACS (acute coronary syndrome) (unstable angina or biomarker positive)
3. Single vessel CAD with at least 2 separate lesions (≥10 mm apart) of ≥40% stenosis or a single long lesion of ≥20mm OR multi-vessel CAD, defined as at least 2 vessels with ≥40% stenosis
4. Pre-PCI iFR performed in all vessels intended for PCI
5. Pre-PCI iFR of <0.90 of at least 1 stenosis
6. Subjects are able and willing to comply with scheduled visits and tests and to provide informed consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant for the duration of the study
2. Acute STEMI (ST-elevated Myocardial Infarction) within the past 7 days
3. Cardiogenic shock (sustained (>10 min) systolic blood pressure < 90 mmHg in absence of inotropic support or the presence of an intra-aortic balloon pump).
4. Ionotropic or temporary pacing requirement
5. Sustained ventricular arrhythmias
6. Prior CABG (Coronary Artery Bypass Graft)
7. Known ejection fraction ≤30%
8. Chronic Total Occlusion (CTO)
9. Known severe mitral or aortic stenosis.
10. Any known medical comorbidity resulting in life expectancy < 12 months.
11. Participation in any investigational study that has not yet reached its primary endpoint.
12. Known severe renal insufficiency (eGFR <30 ml/min/1.72 m2).
13. TIMI flow <3 at baseline
14. Intra-coronary thrombus on baseline angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consented subjects with CAD who undergo physiologic lesion assessment with iFR<0.90 in at least 1 coronary artery are eligible for participation
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Becky Inderbitzen, MSE, Study Director — Philips (Volcano)
Locations (28):
- United States (22):
  - VA Medical Center, Long Beach, California
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Rockford CV Associates, Rockford, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Baystate Medical Center, Springfield, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - South Side Hospital, Bay Shore, New York
  - Northshore Hospital, Manhasset, New York
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - New York Presbyterian Hospital -Weill Cornell, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St Francis Hospital, Roslyn, New York
  - SUNY- Stony Brook, Stony Brook, New York
  - Duke University Hospital, Durham, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Miriam Hospital, Providence, Rhode Island
  - Wellmont CVA Heart Insitute, Kingsport, Tennessee
  - VA North Texas Health Care, Dallas, Texas
  - Aurora St Lukes Medical Center, Milwaukee, Wisconsin
- Netherlands (2):
  - AMC Amsterdam, Amsterdam
  - VU University Medical Center, Amsterdam
- United Kingdom (4):
  - Basildon Univeristy Hospital, Basildon
  - Royal Bournemouth hospital, Bournemouth
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Imperial College of London- Hammersmith Hospital, London

REFERENCES:
- [Result] Jeremias A, Davies JE, Maehara A, Matsumura M, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp A, Ali ZA, Mintz G, Patel M, Stone GW. Blinded Physiological Assessment of Residual Ischemia After Successful Angiographic Percutaneous Coronary Intervention: The DEFINE PCI Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):1991-2001. doi: 10.1016/j.jcin.2019.05.054. PMID 31648761
- [Derived] Patel MR, Jeremias A, Maehara A, Matsumura M, Zhang Z, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp ASP, Ali ZA, Mintz G, Davies J, Stone GW. 1-Year Outcomes of Blinded Physiological Assessment of Residual Ischemia After Successful PCI: DEFINE PCI Trial. JACC Cardiovasc Interv. 2022 Jan 10;15(1):52-61. doi: 10.1016/j.jcin.2021.09.042. PMID 34991824

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI: all participants in the study with analyzable iFR pullback assessment that was performed after a successful PCI, where a successful PCI is assessed based on angiographic results.
Period: Overall Study
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
Started | 500
Analyzable iFR Pullback Assessment Post Angiographically Successful PCI | 467
Completed (completed means study follow-up at 1 year completed) | 463
Not Completed | 37
Not completed — Lost to Follow-up | 32
Not completed — Withdrawal by Subject | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- Diagnostic Test: iFR Pullback: iFR (instantaneous wave free ratio) pullback assessment post angiographically successful PCI
Arm/Group | Diagnostic Test: iFR Pullback
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 379
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (8.8)
Smoker [Count of Participants; unit: Participants] | 83
Diabetes Mellitus [Count of Participants; unit: Participants] | 169
Insulin treated diabetes [Count of Participants; unit: Participants] | 48
Hyperlipidemia [Count of Participants; unit: Participants] | 351
Hypertension [Count of Participants; unit: Participants] | 383
Renal disease [Count of Participants; unit: Participants] | 39
Prior Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 227
Prior Myocardial Infarction [Count of Participants; unit: Participants] | 134
Left ventricular ejection fraction (%) [Mean (Standard Deviation); unit: % of blood ejected with each contraction] | 56.3 (9)
Stable angina [Count of Participants; unit: Participants] | 212
Unstable Angina [Count of Participants; unit: Participants] | 155
NSTEMI (Non-ST Elevated Myocardial Infarction) [Count of Participants; unit: Participants] | 85
Silent Ischemia [Count of Participants; unit: Participants] | 27
Recent STEMI (ST Elevated MI) (>7days) [Count of Participants; unit: Participants] | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Residual Ischemia (iFR <0.90)
Description: Residual ischemia is defined as iFR measurement <0.90 after operator-assessed angiographically successful PCI (residual diameter stenosis <50% in any treated lesion in the target vessel) This outcome describes the number of participants that had a residual ischemia (defined as iFR<0.90) after a PCI that appeared to be successful based on angiography.
Time Frame: end of procedure/intervention
Population: Total vessels/units (535) in participant population (467)
Measure: Number; unit: participants
Units Other Than Participants: Number of vessels in 467 participants
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
Number analyzed (Participants) | 467
Number analyzed (Number of vessels in 467 participants) | 535
participants | 112

2. Secondary Outcome: Cardiac Events
Description: Composite endpoint of cardiac death, target vessel myocardial infarction, ischemia-driven target vessel revascularization or recurrent ischemia at one year after PCI
Time Frame: 12 months
Population: The total number of participants was divided in two groups based on their post-PCI iFR result. (see primary endpoint) The total number of participants still in study at one year is 467.
Measure: Count of Participants; unit: Participants
Groups:
- iFR >= 0.90: Participants with iFR >= 0.90 post-procedure
- iFR < 0.90: Participants with iFR < 0.90 post-procedure
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 9 | 3

3. Secondary Outcome: Target Vessel Failure
Description: Target vessel failure defined as cardiac death, target vessel myocardial infarction, ischemia-driven target vessel revascularization
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 4 | 2

4. Secondary Outcome: Quality of Life Change From Baseline to 12 Months Follow-up
Description: Quality of life (assessed by the Seattle Angina Questionnaire) at baseline, 30-days, 6 months and 1 year (12 months).
  Minimum score is 0 and maximum score is 100, with a high score representing a more positive quality of life score.
  Outcome is the change in score from baseline to 12 months follow-up.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- iFR <= 0.94: post-procedural iFR <= 0.94
- iFR > 0.94: post-procedural iFR > 0.94
Arm/Group | iFR <= 0.94 | iFR > 0.94
Number analyzed (Participants) | 246 | 150
units on a scale | 21.42 (24.99) | 20.73 (21.83)

5. Secondary Outcome: Cardiac Mortality
Description: All-cause and cardiac mortality at one year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 0 | 0

6. Secondary Outcome: Target Vessel MI
Description: Target vessel Myocardial infarction at one year
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 4 | 2

7. Secondary Outcome: Target Vessel Revascularization
Description: Ischemia-driven target vessel revascularization at one year
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 10 | 3

8. Secondary Outcome: Recurrent Ischemia
Description: Recurrent ischemia at one-year
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | iFR >= 0.90 | iFR < 0.90
Number analyzed (Participants) | 355 | 112
Participants | 6 | 1

9. Secondary Outcome: Correlation Between iFR and Angiographic Visual Interpretation
Description: Correlation between iFR <0.90 and coronary stenosis >50% assessed by visual interpretation.
  This was tested using generalized estimating equations for logistic regression to account for the correlation of observations from the same subject.
  An absolute value of exactly 1 implies that a linear equation describes the relationship between iFR and visual interpretation of the angiography.
  Outcome reports how well the iFR value and the visual interpretation are in agreement (for example, when iFR <0.90 and coronary stenosis >50% assessed by visual interpretation the correlation is 1).
Time Frame: at the end of the procedure/intervention
Population: The correlation calculation was performed on the total number of analyzable participants with a post-PCI iFR pullback assessment.
Measure: Number; unit: coefficient of determination (R2)
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
Number analyzed (Participants) | 467
coefficient of determination (R2) | 0.03

10. Secondary Outcome: Number of Participants in Which the iFR Would Become Non-significant if a Focal Stenosis Demonstrated by iFR Pullback Were Treated With PCI
Description: Number of participants in which the iFR would become non-significant if a focal stenosis demonstrated by iFR pullback were treated with PCI
Time Frame: Procedural
Population: This analysis assumes that all focal lesions with post-PCI iFR <0.90 were successfully treated with additional PCI. Using the cutoff of iFR <0.90, the outcome is the number of participants that would remain, or not have been treated, because the iFR measurements are under 0.90.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
Number analyzed (Participants) | 467
Participants | 23

11. Secondary Outcome: Differentiation
Description: Differentiation of the cause for impaired iFR
Time Frame: End of procedure /intervention
Population: Number of vessels in which residual ischemia (post-PCI iFR <0.90) after angiographically successful PCI
Measure: Number; unit: vessels
Units Other Than Participants: vessels
Groups:
- Residual Ischemia (Post-PCI iFR <0.90) After Angiographically Successful PCI: Residual ischemia (post-PCI iFR <0.90)
Arm/Group | Residual Ischemia (Post-PCI iFR <0.90) After Angiographically Successful PCI
Number analyzed (Participants) | 112
Number analyzed (vessels) | 114
vessels
  single or multiple residual focal lesions | 93
  diffuse disease | 21

12. Secondary Outcome: Delta iFR
Description: Predictors of delta iFR before and after PCI, or predictors of impaired iFR Outcome is presented as the odds ratio (OR) that the post-PCI iFR will be <0.90. An OR > 1 means greater odds that the post-PCI iFR is <0.90, OR = 1 means there is no association, and OR < 1 means there is a lower odds that the post-PCI iFR is <0.90.
Time Frame: at the end of the procedure/intervention
Measure: Number; unit: Odds ratio
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
Number analyzed (Participants) | 467
Odds ratio
  pre-PCI reference vessel diameter | 0.32
  lesion location in left anterior descending coronary artery | 5.65

ADVERSE EVENTS:
Time Frame: Adverse Device Effects, Serious Adverse Device Effects, and Unanticipated Adverse Device Effects were collected and if any occurred, they would likely occur during the procedure when the device is being used. Subjects were followed for 12 months and all complaints promptly reported.
Description: As noted above, the only reportable events were Adverse Device Effects, Serious Adverse Device Effects, and Unanticipated Adverse Device Effects.
  Subjects were followed for 12 months, with follow-up visits at 1, 6, and 12 months.
Arm/Group | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI
All-Cause Mortality (participants affected / at risk) | 0/467
Serious Adverse Events (participants affected / at risk) | 12/467
Other Adverse Events (participants affected / at risk) | 0/467
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants With Analyzable iFR Pullback Assessment Post Angiographically Successful PCI (N=467)
Target Vessel Myocardial Infarction (Cardiac disorders) | 6 (6)
Ischemia-driven Target Vessel Revascularization (Cardiac disorders) | 0 (0)
Recurrent Ischemia (Cardiac disorders) | 7 (7)
Cardiac Death (Cardiac disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03084367/Prot_SAP_000.pdf